CLINICAL TRIAL: NCT05763641
Title: Target Axillary Dissection After Neoadjuvant Chemotherapy in Locally Advanced Breast Cancer
Brief Title: TAD After Chemotherapy in Locally Advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, Clinical Professor, Hospital Universitari de Bellvitge
Other Study IDs: PR351/20
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Sentinel Lymph Node; Breast Cancer; Locally Advanced
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Target Axillary Dissection — TAD after neoadjuvant chemotherapy and subsequent axillary lymph node dissection

SUMMARY:
This is an observational study to validate target axillary dissection (TAD) in locally advanced tumors (cN2 and/or cT4).

DETAILED DESCRIPTION:
The procedure will consist of marking the pathological lymph node with 1 clip before the start of neoadjuvant chemotherapy (NAC) and performing surgery after completing the NAC. The TAD will include the exeresis of the node marked with a clip, and of the sentinels marked with technetium and/or patent blue, seeking to obtain at least 3 lymph nodes. Subsequently, the axillary lymphadenectomy will be completed to identify the false negative rate. An initial analysis will be carried out with the first 30 cases, and if there are more than 2 false negative cases, it will be completed until 81 cases of TAD without associated disease are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Axillary lymph node metastasis proven by cytology
* Clinical or radiological N2a (at least 4 suspicious lymph nodes on axillary ultrasound at diagnosis)
* Extensive T4 subsidiary to axillary lymphadenectomy according to current clinical criteria
* Neoadjuvant chemotherapy

Exclusion Criteria:

* cN3 verified by imaging tests
* N2 due to internal mammary involvement (N2b).
* Tumors whose surrogate molecular subtype is luminal A.
* Patients undergoing neoadjuvant endocrine therapy
* Patients with local recurrences and metastatic tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced breast cancer tumours (cN2 or T4) after Neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
TAD validation in locally advanced breast cancer | 3 years
  False negative rate when performing TAD after NAC

SECONDARY OUTCOMES:
Ultrasound validity to evaluate axillary response after NAC | 3 years
  False-negative and positive rates of axillary ultrasound after NAC to assess lymph node response
MRI validity to evaluate axillary response after NAC | 3 years
  False-negative and positive rates of axillary MRI after NAC to asses lymph node response

CONTACTS AND LOCATIONS:
Overall Officials: amparo Garcia-Tejedor, MDPhD, Principal Investigator — Instituto de Investigación Biomédica de Bellvitge (IDIBELL)
Locations (2):
- Spain (2):
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided